CLINICAL TRIAL: NCT06621134
Title: Comparing the Effectiveness of an AI Chatbot with That of a Telephone Hotline for Answering COVID-19 Related Issues
Brief Title: Comparing the Effectiveness of AI Chatbot with That of Telephone Hotline
Acronym: AI chatbot
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Patrick Ip, Clinical Professor, The University of Hong Kong
Other Study IDs: UW21-344; Collaborative Research Fund (Other Grant/Funding Number: University Grants Committee)
Record Dates: First submitted 2024-09-16; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Telephone Hotlines; AI Chatbot
Keywords: Artificial Intelligence; AI chatbot
MeSH Terms: interventions — Hotlines

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control Group: Participants will be asked to consent to randomization on their first access to our system. Users ask questions covered by the question bank and specific questions not covered by the question through a telephone hotline.
  Interventions: Other: Telephone hotline
- Intervention Group: Participants will be required to provide consent for randomization when they first access our system. Users can ask questions covered by the question bank, as well as specific questions not covered by the bank, through an AI chatbox.
  Interventions: Other: AI Chatbot

INTERVENTIONS:
Other: AI Chatbot — Participants will be required to provide consent for randomization when they first access our system. Users can ask questions covered by the question bank, as well as specific questions not covered by the bank, through an AI chatbox. The aim is to understand the significant difference between using AI chatbots and telephone hotlines to assist parents, as well as the effectiveness of AI chatbots compared to telephone hotlines.
  Groups: Intervention Group
Other: Telephone hotline — Participants will be asked to consent to randomization on their first access to our system. Users ask questions covered by the question bank and specific questions not covered by the question through a telephone hotline.
  Groups: Control Group

SUMMARY:
The COVID-19 pandemic has significantly impacted the wellbeing of people in Hong Kong, leading to social distancing policies and changes in healthcare service utilization. School closures and remote work have increased stress levels for parents and children. Vulnerable populations, such as low-income families and children with special needs, are at higher risk of maltreatment and mental health issues. Parental burnout has become a concern as parents juggle work, childcare, and education responsibilities. There is a need for research on the physical and mental health effects of COVID-19 on families and the potential role of AI in addressing these challenges. AI, particularly chatbots, can provide accessible healthcare information and support, aiding in early diagnosis and treatment. AI chatbots offer timely responses, accurate information, and continuous availability, making them valuable tools for remote health assistance. While AI chatbots are not without limitations, further research can help integrate them more effectively into healthcare services.

DETAILED DESCRIPTION:
The COVID-19 pandemic has had an unprecedented impact on the wellbeing of people in Hong Kong since the outbreak in December 2019. The Government has adopted social distancing policies to minimise the risk of infection. These include but are not limited to; school closure, remote working, and the prohibition of group-gatherings. These anti-infection measures have led to a change in pattern in the use of healthcare services and help-seeking activities. Studies have also shown that a dearth of socialisation leads to higher stress levels for both parents and children.

As school closure and remote work measures continue, both children and parents are under great pressure. UNESCO (2020) reported that over 1.58 billion children and youth in 200 countries were affected by school closure, as of mid-April 2020. Although the long-term effect of COVID-19 on children's and parents' mental health is unknown, cases of child abuse, neglect and exploitation have increased in the face of such unprecedented times. Low-income families or families with children with special education needs (SEN) are prone to children being maltreated and/or having mental health crisis . Parents who work from home are facing challenges of fulfilling a triple role: work, childcare and homecare. Worse still, children's lack of learning interests and motivation adds extra burden on parents as they take up the role of teachers. Parents are inclined to experience parental burnout, which is characterised by mental and physical exhaustion, with a feeling of hopelessness. Therefore it is clear there are strong societal needs for COVID-19 physical and mental health research. It is imperative to prevent potential and mitigate existing problems regarding parent-child relationship, parental stress and family functioning caused by COVID-19.

Consequently, exploring more easily accessible and efficient ways of dealing with potential and existing health problems (both physically and mentally) should be a priority. Artificial Intelligence (AI) in healthcare services has the potential to reduce the workload of healthcare workers by answering frequently asked questions through the AI system all from the comfort of the subject's home. Considering the potentially detrimental effect of COVID-19 on both children and parents it is important to fill the research gap as to how AI may serve as a platform for help-seeking, particularly during times of social distancing.

AI has been widely adopted in healthcare services in the past decade. The use of chatbots, in particular, has enhanced public engagement in health service all from the comfort of the subject's home. AI chatbots utilised natural language processing (NLP) to facilitate interaction with users in conversations, making appropriate medical advice accessible to the public. Intelligent algorithms in AI enables early diagnosis of disease and offers treatment techniques to those who may otherwise have been diagnosed too late. For instance, the U.S. Centres for Disease Control and Prevention (CDC) has launched a chatbot named Clara to help users access information on potential symptoms of coronavirus and help enable them to make decisions about the need to seek medical care). This is especially useful as it identifies high-risks groups in need of medical attention by triaging patients according to their symptoms, therefore reducing hospital visits for minor cases. It also provides support to family members of high-risk groups as to what measures can be taken to prevent infection and ways to relieve pressure in taking care of patients within their family.

AI chatbots merit attention in its prompt response to users' questions as it provides a service around the clock. In addition, answers provided by AI are considered more accurate than that of search engines, subject to the proficiency of data mining methods. These features are of significance as users are able to seek psycho-medical advice while practising social distancing, without face-to-face appointments with clinicians.

AI chatbots may serve as a self-help tool for gaining insights in dealing with both mental and physical conditions but it is far from perfection. The hope is that this study can contribute to making AI chatbots an integrated part of the health care service.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who give consent to participate in the study.

Exclusion Criteria:

* Subjects who do not give consent to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: No specific population
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2021-09-03 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
General Anxiety Disorder (GAD - 7) | 1 week within Pre-test, 1 week within Post-test
  The Generalized Anxiety Disorder 7-item (GAD-7) questionnaire is a self-reported screening tool used to assess the severity of generalized anxiety disorder symptoms in adults. It consists of seven questions that ask about various symptoms commonly associated with generalized anxiety disorder, such as feeling nervous, anxious, or on edge.General Anxiety Disorder (GAD - 7)
Patient Health Questionnaire-9 | 1 week within Pre-test, 1 week within Post-test
  The Patient Health Questionnaire-9 (PHQ-9) is a self-administered questionnaire used to screen for and assess the severity of depression in patients. It consists of nine questions based on the criteria for diagnosing major depressive disorder in the Diagnostic and Statistical Manual of Mental Disorders (DSM-5). Patients are asked to rate how often they have experienced certain symptoms of depression over the past two weeks, with response options ranging from "not at all" to "nearly every day." The total score on the PHQ-9 can help healthcare providers determine the presence and severity of depression in a patient, as well as monitor their response to treatment over time.

SECONDARY OUTCOMES:
Service Satisfaction Survey | 1 week within Pre-test, 1 week within Post-test
  A Service Satisfaction Survey is a method used by organizations to collect feedback from customers or clients regarding their satisfaction with the services provided. These surveys typically include questions that assess various aspects of the service experience, such as quality, responsiveness, professionalism, and overall satisfaction. The feedback gathered from these surveys can help organizations identify areas for improvement and make informed decisions to enhance their services.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Paediatrics and Adolescent Medicine, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tso WWY, Wong RS, Tung KTS, Rao N, Fu KW, Yam JCS, Chua GT, Chen EYH, Lee TMC, Chan SKW, Wong WHS, Xiong X, Chui CS, Li X, Wong K, Leung C, Tsang SKM, Chan GCF, Tam PKH, Chan KL, Kwan MYW, Ho MHK, Chow CB, Wong ICK, Lp P. Vulnerability and resilience in children during the COVID-19 pandemic. Eur Child Adolesc Psychiatry. 2022 Jan;31(1):161-176. doi: 10.1007/s00787-020-01680-8. Epub 2020 Nov 17. PMID 33205284
- [Background] Russell BS, Hutchison M, Tambling R, Tomkunas AJ, Horton AL. Initial Challenges of Caregiving During COVID-19: Caregiver Burden, Mental Health, and the Parent-Child Relationship. Child Psychiatry Hum Dev. 2020 Oct;51(5):671-682. doi: 10.1007/s10578-020-01037-x. PMID 32749568
- [Background] Naseem M, Akhund R, Arshad H, Ibrahim MT. Exploring the Potential of Artificial Intelligence and Machine Learning to Combat COVID-19 and Existing Opportunities for LMIC: A Scoping Review. J Prim Care Community Health. 2020 Jan-Dec;11:2150132720963634. doi: 10.1177/2150132720963634. PMID 32996368
- [Background] Lee J. Mental health effects of school closures during COVID-19. Lancet Child Adolesc Health. 2020 Jun;4(6):421. doi: 10.1016/S2352-4642(20)30109-7. Epub 2020 Apr 14. No abstract available. PMID 32302537
- [Background] Kretzschmar K, Tyroll H, Pavarini G, Manzini A, Singh I; NeurOx Young People's Advisory Group. Can Your Phone Be Your Therapist? Young People's Ethical Perspectives on the Use of Fully Automated Conversational Agents (Chatbots) in Mental Health Support. Biomed Inform Insights. 2019 Mar 5;11:1178222619829083. doi: 10.1177/1178222619829083. eCollection 2019. PMID 30858710
- [Background] Garrido S, Millington C, Cheers D, Boydell K, Schubert E, Meade T, Nguyen QV. What Works and What Doesn't Work? A Systematic Review of Digital Mental Health Interventions for Depression and Anxiety in Young People. Front Psychiatry. 2019 Nov 13;10:759. doi: 10.3389/fpsyt.2019.00759. eCollection 2019. PMID 31798468
- [Background] Cluver L, Lachman JM, Sherr L, Wessels I, Krug E, Rakotomalala S, Blight S, Hillis S, Bachman G, Green O, Butchart A, Tomlinson M, Ward CL, Doubt J, McDonald K. Parenting in a time of COVID-19. Lancet. 2020 Apr 11;395(10231):e64. doi: 10.1016/S0140-6736(20)30736-4. Epub 2020 Mar 25. No abstract available. PMID 32220657
- [Background] Chew AMK, Ong R, Lei HH, Rajendram M, K V G, Verma SK, Fung DSS, Leong JJ, Gunasekeran DV. Digital Health Solutions for Mental Health Disorders During COVID-19. Front Psychiatry. 2020 Sep 9;11:582007. doi: 10.3389/fpsyt.2020.582007. eCollection 2020. No abstract available. PMID 33033487
- See also: Nature — https://www.nature.com/articles/npjschz201530
- See also: Global economic observer — https://ideas.repec.org/a/ntu/ntugeo/vol6-iss2-18-071.html
- See also: HKSAR Government — https://www.info.gov.hk/gia/general/202012/08/P2020120800780.htm